CLINICAL TRIAL: NCT01689467
Title: Efficacy and Safety of Fermented Velvet Antler Extract on Fatigue Recovery After Exercise
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chonbuk National University Hospital (Other)
Responsible Party: Principal Investigator, Soo-Wan Chae, Clinical Trial Center for Functional Foods, Chonbuk National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: KD-FR-FVE
Record Dates: First submitted 2012-09-18; First posted 2012-09-21 (Estimated); Last update posted 2019-08-26 (Actual); Status verified 2019-08

CONDITIONS: Chronic Fatigue Syndrome
MeSH Terms: conditions — Fatigue Syndrome, Chronic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Fermented Velvet Antler extract (Experimental)
  Interventions: Dietary Supplement: Fermented Velvet Antler extract
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Fermented Velvet Antler extract — Fermented Velvet Antler extract (1g/day)
  Arms: Fermented Velvet Antler extract
Dietary Supplement: Placebo — Placebo (1g/day)
  Arms: Placebo

SUMMARY:
The investigators performed a 12-week, randomized, double-blind, placebo-controlled human trial to evaluate the efficacy and safety of Fermented Velvet Antler extract on fatigue recovery after exercise. The investigators measured fatigue recovery parameters , including lactate, ammonia, inorganic phosphorus, creatine kinase and LDH, and monitored their blood pressure.

ELIGIBILITY:
Inclusion Criteria:

* Males and females 19-60 years old
* Hemoglobin concentration between 13 and 14 g/dL(men), 12 and 13 g/dL(women)
* Able to give informed consent

Exclusion Criteria:

* Allergic or hypersensitive to any of the ingredients in the test products
* History of reaction to any of the test products or of gastrointestinal diseases such as Crohn's disease or gastrointestinal surgery
* Participation in any other clinical trials within past 2 months
* Laboratory test, medical or psychological conditions deemed by the investigators to interfere with successful participation in the study
* Pregnant or lactating women etc.

Ages: 19 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2013-04-25 (Actual); Primary Completion 2014-06-26 (Actual); Study Completion 2014-06-26 (Actual)

PRIMARY OUTCOMES:
Changes in lactate | 12 weeks
  Lactate was measured in study visit 1(0 week) and visit 3(12 week).
Changes in ammonia | 12 weeks
  Ammonia was measured in study visit 1(0 week) and visit 3(12 week).
Changes in inorganic phosphorus | 12 weeks
  Inorganic phosphorus was measured in study visit 1(0 week) and visit 3(12 week).
Changes in creatine kinase | 12 weeks
  Creatine kinase was measured in study visit 1(0 week) and visit 3(12 week).
Changes in Lactage dehydrogenase(LDH) | 12 weeks
  Lactage dehydrogenase(LDH) was measured in study visit 1(0 week) and visit 3(12 week).

SECONDARY OUTCOMES:
Changes in Multidimensional Fatigue Scale(MFS) | 12 weeks
  Multidimensional Fatigue Scale(MFS) was measured in study visit 1(0 week) and visit 3(12 week).
Changes in 36-Item Short-Form Health Survey(SF-36) | 12 weeks
  36-Item Short-Form Health Survey(SF-36) was measured in study visit 1(0 week) and visit 3(12 week).

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Trial Center for Functional Foods; Chonbuk National University Hospital, Jeonju, Jeollabuk-do, South Korea